CLINICAL TRIAL: NCT01665937
Title: A Phase I Study of STA-9090 in Patients With Advanced Hepatocellular Carcinoma
Brief Title: STA-9090 in Patients With Advanced Hepatocellular Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Beth Israel Deaconess Medical Center (Other); Synta Pharmaceuticals Corp. (Industry)
Responsible Party: Principal Investigator, Andrew X. Zhu, MD, MD, PhD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-072
Record Dates: First submitted 2010-04-27; First posted 2012-08-16 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: liver cancer; advanced liver cancer; advanced hepatocellular cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — STA 9090

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- STA-9090 (Experimental): Patients receiving STA-9090
  Interventions: Drug: STA-9090

INTERVENTIONS:
Drug: STA-9090 — IV one time weekly for 3 weeks in 4 week cycles. Study treatment is given in 4-week time periods called cycles. Patients will receive STA-9090 for the first 3 weeks of each cycle and no treatment on the fourth week. STA-9090 will be given by intravenous (IV) infusion. IV infusions occur through an IV catheter (or tube) placed in the vein. Each infusion will last about 60 minutes.
  During each cycles patients will have blood tests, pregnancy test, and EKG. Twenty to thirty days after the last dose, patients will return for a physical exam, blood tests, urine test, EKG, and CT or MRI of chest and abdomen.

SUMMARY:
STA-9090 works by inhibiting the function of a protein in tumor cells called Hsp90. Hsp90 is thought to play a role in tumor growth. By interfering with this protein's function, STA-9090 may help kill tumor cells. This drug has been used in other research studies and information from those studies suggests that this agent may help to slow tumor growth in HCC.

The purpose of this research study is to find the highest dose of STA-9090 that can safely be given to participants with advanced HCC. The investigators will also get more information about the safety of STA-9090 and perform tests to learn more about how STA-9090 affects the body.

DETAILED DESCRIPTION:
Study treatment is given in 4-week time periods called cycles. Patients will receive ST-9090 once weekly for the first 3 weeks of each cycle and no treatment on the fourth week. STA-9090 will be given by intravenous (IV) infusion. IV infusions occur through an IV catheter (or tube) placed in the vein. Each infusion will last about 60 minutes.

During each cycles patients will have blood tests, pregnancy test, and EKG. Twenty to thirty days after the last dose, patients will return for a physical exam, blood tests, urine test, EKG, and CT or MRI of chest and abdomen.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed hepatocellular carcinoma
* Measurable disease
* Life expectancy greater than 3 months
* ECOG performance status 0 or 1
* BCLC Stage C disease
* Lab values must be within limits outlined in protocol
* Child-Pugh score </= 6
* CLIP score 0-3
* Must agree to use adequate contraception

Exclusion Criteria:

* Chemotherapy or radiotherapy within 4 weeks prior to entering study or not recovered from adverse events due to agents administered more than 4 weeks earlier
* Receiving any other investigational agent
* Known brain metastases unless treated and radiographically and clinically stable without steroid or anticonvulsant medications for at least 4 weeks prior to first dose of STA-9090
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to STA-9090
* Surgery, radiotherapy, or lesion ablative procedure to the only area of measurable disease
* Major surgery within 4 weeks prior to first dose of STA-9090
* Poor venous access for study drug administration or would require a peripheral or central indwelling catheter for study drug administration
* History of severe allergic or hypersensitivity reactions to excipients (e.g., Polyethylene glycol [PE] 300 and Polysorbate 80)
* Baseline QTc > 450 msec or previous history of QT prolongation while taking other medications
* Ventricular ejection fraction </= 55% at baseline
* Treatment with chronic immunosuppressants
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breast-feeding
* History of a different malignancy unless disease-free for at least 5 years and deemed by the investigator to be at low risk for recurrence.
* HIV-positive individuals on combination antiretroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-08; Primary Completion 2013-07 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Phase 2 dose of STA 9090 given once weekly in patients with advanced hepatocellular carcinoma | 3 years
  Dose escalation/de-escalation study will be performed in order to determine the Phase 2 dose of STA-9090 given once weekly in patients with advanced hepatocellular carcinoma. The dose limiting toxicities will be determined at each dose level.

SECONDARY OUTCOMES:
Number of patients with adverse events when treated with STA 9090 for advanced hepatocellular carcinoma | 3 years
  To assess the safety and tolerability of STA9090 in patients with advanced hepatocellular carcinoma.
Median time to progression (TTP) | 3 years
  To determine median time to progression (TTP) for patients treated at recommended Phase 2 dose.
Median progression-free survival (PFS) | 3 years
  To determine median progression-free survival (PFS) for patients treated at recommended Phase 2 dose.
Response Rate | 3 years
  To determine objective tumor response rate using RECIST criteria
Overall Survival | 3 years
  To determine overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Zhu, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No